CLINICAL TRIAL: NCT03266016
Title: Identifying and Preventing Ventilator Induced Diaphragm Dysfunction in Children
Brief Title: Real-time Effort Driven VENTilator Management
Acronym: REDvent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Robinder Khemani, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHLA-17-00235; 5R01HL134666-05 (NIH)
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Ventilation Therapy; Complications; Diaphragm Disease; Pediatric Respiratory Diseases
MeSH Terms: interventions — Maximal Respiratory Pressures

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Analysis Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- REDvent-acute (Experimental): Acute Phase: The acute phase is defined as the time from intubation until the patient meets weaning criteria, passes the initial oxygenation test (decrease PEEP to 5 cmH2O and FiO2 to 0.5, maintains SpO2 > 90%), and undergoes a Spontaneous Breathing Trial (SBT). Patients will be managed with pressure control plus pressure support ventilation using a computerized decision support tool that will recommend changes to ventilator settings approximately every 4 hr (with or without a new blood gas). If the patient is spontaneously breathing, it will incorporate real-time measures of effort of breathing (esophageal manometry) to keep it in a target range.
  Interventions: Other: Computerized Ventilator Protocol; Diagnostic Test: Esophageal Manometry; Diagnostic Test: Respiratory Inductance Plethysmography (RIP); Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Maximal Inspiratory Pressure
- Control-acute (Placebo Comparator): Acute Phase: The acute phase is defined as the time from intubation until the patient meets weaning criteria, passes the initial oxygenation test (decrease PEEP to 5 cmH2O and FiO2 to 0.5, maintains SpO2 > 90%), and undergoes a Spontaneous Breathing Trial (SBT). Ventilator management will be per usual care until the patient meets weaning criteria and passes the oxygenation test.
  Interventions: Diagnostic Test: Esophageal Manometry; Diagnostic Test: Respiratory Inductance Plethysmography (RIP); Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Maximal Inspiratory Pressure
- REDvent-weaning (Experimental): Weaning Phase: The weaning phase is defined as the time from the first Spontaneous Breathing Trial (SBT) until the patient successfully passes an SBT or is extubated (whichever comes first). Patients who pass the initial SBT at the end of the acute phase will not undergo weaning phase randomization. Patients will be managed in a pressure support/CPAP mode of ventilation with assessments or changes to the level of pressure support every 4 hours, targeting maintaining effort of breathing (esophageal manometry) in a normal range. An SBT will be conducted daily, and the weaning phase will continue until the patient passes the SBT.
  Interventions: Other: Computerized Ventilator Protocol; Diagnostic Test: Esophageal Manometry; Diagnostic Test: Respiratory Inductance Plethysmography (RIP); Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Maximal Inspiratory Pressure
- Control-weaning (Placebo Comparator): Weaning Phase: The weaning phase is defined as the time from the first Spontaneous Breathing Trial (SBT) until the patient successfully passes an SBT or is extubated (whichever comes first). Patients who pass the initial SBT at the end of the acute phase will not undergo weaning phase randomization. Ventilator management will be per usual care. An SBT will be conducted daily, and the weaning phase will continue until the patient passes the SBT.
  Interventions: Diagnostic Test: Esophageal Manometry; Diagnostic Test: Respiratory Inductance Plethysmography (RIP); Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Maximal Inspiratory Pressure

INTERVENTIONS:
Other: Computerized Ventilator Protocol — Computerized Decision Support System which recommends changes to ventilator settings to promote physiologic levels of patient effort of breathing.
  Arms: REDvent-acute; REDvent-weaning
Diagnostic Test: Esophageal Manometry — Esophageal Manometry Catheter to measure effort of breathing an transpulmonary pressure
Diagnostic Test: Respiratory Inductance Plethysmography (RIP) — RIP bands to measure thoraco-abdominal synchrony during spontaneous breathing trials
Diagnostic Test: Diaphragm Ultrasound — Daily measurement of diaphragm thickness and diaphragm contractile activity
Diagnostic Test: Maximal Inspiratory Pressure — Prior to Spontaneous breathing trials, measurement of airway and esophageal maximal inspiratory pressure during airway occlusion

SUMMARY:
This study is a Phase II controlled clinical trial that will obtain comprehensive, serial assessments of respiratory muscle strength and architecture to understand the evolution of ventilator-induced respiratory muscle weakness in critically ill children, and test whether a novel computer-based approach (Real-time Effort Driven ventilator management (REDvent)) can preserve respiratory muscle strength and reduce time on MV. REDvent offers systematic recommendations to reduce controlled ventilation during the acute phase of MV, and uses real-time measures from esophageal manometry to adjust supported ventilator pressures such that patient effort of breathing remains in a normal range during the ventilator weaning phase. This phase II clinical trial is expected to enroll 276 children with pulmonary parenchymal disease, anticipated to be ventilated > 48 hrs. Patients will be randomized to REDvent-acute vs. usual care for the acute phase of MV (interval from intubation to first spontaneous breathing trial (SBT)). Patients in either group who fail their first Spontaneous Breathing Trial (SBT), will also be randomized to REDvent-weaning vs. usual care for the weaning phase of MV (interval from first SBT to passing SBT). The primary clinical outcome is length of weaning (time from first SBT until successful passage of an SBT or extubation (whichever comes first)). Mechanistic outcomes surround multi-modal serial measures of respiratory muscle capacity (PiMax), load (resistance, compliance), effort (esophageal manometry), and architecture (ultrasound) throughout the course of MV. Upon completion, this study will provide important information on the pathogenesis and timing of respiratory muscle weakness during MV in children and whether this weakness can be mitigated by promoting more normal patient effort during MV via the use of REDvent. This will form the basis for a larger, Phase III multi-center study, powered for key clinical outcomes such as 28-day Ventilator Free Days.

DETAILED DESCRIPTION:
Study Aims:

SA1: To determine if REDvent acute and/or weaning phase protocols can shorten the duration of weaning from MV (Primary outcome).

SA2: To determine if changes to direct measures of respiratory muscle strength, load, effort, and architecture throughout the duration of MV are related to weaning outcomes.

SA3: To determine if patient effort of breathing during both acute and weaning phases of MV is independently associated with the development of respiratory muscle weakness.

Study Design: Single-center randomized controlled trial (138 children per arm) using REDvent (intervention arm) as compared with usual care ventilator management including a standardized daily SBT (control arm). Acute phase randomization will occur upon study enrollment, and patients who fail the first SBT will undergo a weaning phase randomization. The investigators will obtain serial measurements of respiratory system capacity, load, effort of breathing, and diaphragm architecture throughout the course of MV.

Acute Phase: The acute phase is defined as the time from intubation until the patient meets weaning criteria, passes the initial oxygenation test (decrease PEEP to 5 cmH2O and FiO2 to 0.5, maintains SpO2 > 90%), and undergoes a Spontaneous Breathing Trial (SBT).

1. Intervention Arm (REDvent-acute): Patients will be managed with pressure control plus pressure support ventilation using a computerized decision support tool that will recommend changes to ventilator settings approximately every 4 hr (with or without a new blood gas). If the patient is spontaneously breathing, it will incorporate real-time measures of effort of breathing (esophageal manometry) to keep it in a target range.
2. Control Arm (Control-acute): Ventilator management will be per usual care until the patient meets weaning criteria and passes the oxygenation test.

Weaning Phase: The weaning phase is defined as the time from the first Spontaneous Breathing Trial (SBT) until the patient successfully passes an SBT or is extubated (whichever comes first). Patients who pass the initial SBT at the end of the acute phase will not undergo weaning phase randomization.

1. Intervention Arm (REDvent-weaning): Patients will be managed in a pressure support/CPAP mode of ventilation with assessments or changes to the level of pressure support every 4 hours, targeting maintaining effort of breathing (esophageal manometry) in a normal range. An SBT will be conducted daily, and the weaning phase will continue until the patient passes the SBT.
2. Control Arm (Control-weaning): Ventilator management will be per usual care. An SBT will be conducted daily, and the weaning phase will continue until the patient passes the SBT.

Analysis Plan and Sample Size Justification:

Aim 1: The primary outcome is weaning duration. Sample size has been determined to adequately power 3 separate comparative analyses: (a) REDvent-acute versus Acute Phase control (b) REDvent-weaning phase versus Weaning Phase control (c) REDvent both phases versus control both phases. Power is based on 2 planned methods for analysis: cox proportional hazard ratios for multivariable analysis and univariate analysis with an independent t-test using log transformation (as needed) to account for the expected distribution of weaning duration. For all three of the planned comparisons above, with the proposed sample size the investigators would be adequately powered (>0.8) to detect a difference in weaning duration of ≥ 1 day, or a hazard ratio of ≥ 1.4 between groups. The secondary outcomes are ventilator free days and extubation failure. Directly comparing control only patients to REDvent only patients, with an expected standard deviation for VFDs between 5 to 9 days, the investigators will be able to detect a 2-day change in VFDs between groups with a power between 0.35 and 0.82. Re-intubation rates are expected to be 10%, allowing the investigators to confirm that REDvent is not inferior to usual care in regards to re-intubation with a non-inferiority margin of 0.10 with a power of 0.8 and alpha of 0.05.

Aim 2: The primary outcome of this aim is weaning duration. For respiratory muscle strength the investigators will compare the first measured aPiMax (after resolution of the acute phase, before the first SBT), the trajectory and value of the daily aPiMax during the weaning phase prior to extubation, the lowest and highest measured aPiMax, and aPiMax on the day of extubation against weaning duration. For analysis, aPiMax will be dichotomized at 30 cmH2O, and weaning duration will be compared between patients with aPiMax > 30 versus ≤ 30 cmH2O using a t-test with or without log-transformation, or Mann-Whitney U test, depending on the distribution. From preliminary data, it is anticipated at least 35% of patients (n=84) will have aPiMax ≤ 30 cmH2O. Based on a similar power analysis as presented above, this would allow the investigators to determine whether low aPiMax is associated with a ≥ 1-day increase in weaning duration, with an alpha of 0.05 and power of 0.8. The investigators will perform identical analysis for ePiMax. Diaphragm Thickness analysis will compound daily ultrasound measures to detect the relative change in diaphragm thickness from study day 1 until passage of an SBT. The investigators will compare the change in thickness after resolution of the acute phase (on the day of the first SBT) against weaning duration, in a similar manner as proposed above for aPiMax. In addition to weaning duration, the investigators will also examine whether the respiratory measures taken just prior to or during each SBT are associated with the patient passing the SBT. For example with aPiMax and ePiMax, the investigators will examine if there is a dose response relationship between PiMax measured just before the SBT and the rate of passage of the subsequent SBT.

Aim 3: The primary outcome of this aim is aPiMax < 30 cmH2O.The analysis will focus on determining whether the degree of patient effort of breathing is independently associated with the development of respiratory muscle weakness. For the acute phase, the investigators will generate a time-weighted average PRP during the acute phase and graph it against aPiMax at the first SBT. They will subsequently dichotomize aPiMax at the first SBT and compare mean time weighted average PRP in the acute phase between aPiMax groups (> 30 vs. ≤ 30 cmH2O). For the weaning phase, the investigators will graph the changes in aPiMax throughout the weaning phase (from first failed SBT until successful SBT) against time-weighted average PRP, with the anticipation that low PRP will be associated with either further reductions in aPiMax, or no improvement, while PRP in the physiologic range of 150-400 will be associated with improvement in aPiMax. The investigators will subsequently dichotomize aPiMax (at 30 cm H2O) at the time of successful passage of an SBT and compare time-weighted average PRP in the weaning phase between aPiMax groups. Subsequently, the investigators will build a multivariable logistic regression model on the outcome of aPiMax ≤ 30 cmH2O to determine if time-weighted PRP in the acute phase, weaning phase or both have an independent association with preserving aPiMax, after controlling for confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Children > 1 month (>44 weeks CGA) and ≤ 18 years of age AND
* Supported on mechanical ventilation with pulmonary parenchymal disease (i.e., pneumonia, bronchiolitis, Pediatric Acute Respiratory Distress Syndrome (PARDS)) with Oxygen Saturation Index (OSI) ≥ 5 or Oxygenation Index (OI) ≥) AND
* Who are within 48 hours of initiation of invasive mechanical ventilation (allow for up to 72 hours for those transferred from another institution)

Exclusion Criteria:

* Contraindications to use of an esophageal catheter (i.e. severe mucosal bleeding, nasal encephalocele, transphenoidal surgery) OR
* Contraindications to use of RIP bands (i.e. omphalocele, chest immobilizer or cast) OR
* Conditions precluding diaphragm ultrasound measurement (i.e. abdominal wall defects, pregnancy) OR
* Conditions on enrollment that preclude conventional methods of weaning (i.e., status asthmaticus, severe lower airway obstruction, critical airway, intracranial hypertension, Extra Corporeal Life Support (ECLS), intubation for UAO, DNR, severe chronic respiratory failure, spinal cord injury above lumbar region, cyanotic heart disease (unrepaired or palliated)) OR
* Primary Attending physician refuses (will be cleared with primary attending before approaching the patient).

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 248 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robinder G Khemani, MD, MsCI, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified IPD will be made available as per NIH guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: Within 5 years of publication of primary manuscript
Access Criteria: Will be made available through biolinc
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Derived] Khemani RG, Bhalla A, Hotz JC, Klein MJ, Kwok J, Kohler K, Bornstein D, Chang D, Armenta-Quiroz A, Vu K, Smith E, Suresh A, Baron D, Bonilla-Cartagena J, Ross PA, Deakers T, Beltramo F, Nelson L, Shah S, Elkunovich M, Curley MAQ, Mack W, Newth CJL. Randomized Trial of Lung and Diaphragm Protective Ventilation in Children. NEJM Evid. 2025 Jun;4(6):EVIDoa2400360. doi: 10.1056/EVIDoa2400360. Epub 2025 May 27. PMID 40423397
- [Derived] Vedrenne-Cloquet M, Ito Y, Hotz J, Klein MJ, Herrera M, Chang D, Bhalla AK, Newth CJL, Khemani RG. Phenotypes based on respiratory drive and effort to identify the risk factors when P0.1 fails to estimate ∆PES in ventilated children. Crit Care. 2024 Oct 4;28(1):325. doi: 10.1186/s13054-024-05103-x. PMID 39367452
- [Derived] Ito Y, Herrera MG, Hotz JC, Kyogoku M, Newth CJL, Bhalla AK, Takeuchi M, Khemani RG. Estimation of inspiratory effort using airway occlusion maneuvers in ventilated children: a secondary analysis of an ongoing randomized trial testing a lung and diaphragm protective ventilation strategy. Crit Care. 2023 Nov 29;27(1):466. doi: 10.1186/s13054-023-04754-6. PMID 38031116
- [Derived] Knox KE, Hotz JC, Newth CJL, Khoo MCK, Khemani RG. A 30-Minute Spontaneous Breathing Trial Misses Many Children Who Go On to Fail a 120-Minute Spontaneous Breathing Trial. Chest. 2023 Jan;163(1):115-127. doi: 10.1016/j.chest.2022.08.2212. Epub 2022 Aug 28. PMID 36037984
- [Derived] van Dijk J, Blokpoel RGT, Abu-Sultaneh S, Newth CJL, Khemani RG, Kneyber MCJ. Clinical Challenges in Pediatric Ventilation Liberation: A Meta-Narrative Review. Pediatr Crit Care Med. 2022 Dec 1;23(12):999-1008. doi: 10.1097/PCC.0000000000003025. Epub 2022 Jul 14. PMID 35830707
- [Derived] Shimatani T, Yoon B, Kyogoku M, Kyo M, Ohshimo S, Newth CJL, Hotz JC, Shime N, Khemani RG. Frequency and Risk Factors for Reverse Triggering in Pediatric Acute Respiratory Distress Syndrome during Synchronized Intermittent Mandatory Ventilation. Ann Am Thorac Soc. 2021 May;18(5):820-829. doi: 10.1513/AnnalsATS.202008-1072OC. PMID 33326335
- [Derived] Khemani RG, Hotz JC, Klein MJ, Kwok J, Park C, Lane C, Smith E, Kohler K, Suresh A, Bornstein D, Elkunovich M, Ross PA, Deakers T, Beltramo F, Nelson L, Shah S, Bhalla A, Curley MAQ, Newth CJL. A Phase II randomized controlled trial for lung and diaphragm protective ventilation (Real-time Effort Driven VENTilator management). Contemp Clin Trials. 2020 Jan;88:105893. doi: 10.1016/j.cct.2019.105893. Epub 2019 Nov 16. PMID 31740425

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute: REDvent: Acute Phase: The acute phase is defined as the time from intubation until the patient meets weaning criteria, passes the initial oxygenation test (decrease PEEP to 5 cmH2O and FiO2 to 0.5, maintains SpO2 > 90%), and undergoes a Spontaneous Breathing Trial (SBT). Patients will be managed with pressure control plus pressure support ventilation using a computerized decision support tool that will recommend changes to ventilator settings approximately every 4 hr (with or without a new blood gas). If the patient is spontaneously breathing, it will incorporate real-time measures of effort of breathing (esophageal manometry) to keep it in a target range.
  Computerized Ventilator Protocol: Computerized Decision Support System which recommends changes to ventilator settings to promote physiologic levels of patient effort of breathing.
  Esophageal Manometry: Esophageal Manometry Catheter to measure effort of breathing an transpulmonary pressure
  Respiratory Inductance Plethysmography (RIP): RIP bands to measure thoraco-abdominal synchrony during spontaneous breathing trials
  Diaphragm Ultrasound: Daily measurement of diaphragm thickness and diaphragm contractile activity
  Maximal Inspiratory Pressure: Prior to Spontaneous breathing trials, measurement of airway and esophageal maximal inspiratory pressure during airway occlusion
- Acute: Control: Acute Phase: The acute phase is defined as the time from intubation until the patient meets weaning criteria, passes the initial oxygenation test (decrease PEEP to 5 cmH2O and FiO2 to 0.5, maintains SpO2 > 90%), and undergoes a Spontaneous Breathing Trial (SBT). Ventilator management will be per usual care until the patient meets weaning criteria and passes the oxygenation test.
  Esophageal Manometry: Esophageal Manometry Catheter to measure effort of breathing an transpulmonary pressure
  Respiratory Inductance Plethysmography (RIP): RIP bands to measure thoraco-abdominal synchrony during spontaneous breathing trials
  Diaphragm Ultrasound: Daily measurement of diaphragm thickness and diaphragm contractile activity
  Maximal Inspiratory Pressure: Prior to Spontaneous breathing trials, measurement of airway and esophageal maximal inspiratory pressure during airway occlusion
- Weaning: Redvent: The weaning phase is defined as the time from the first SBT until the patient successfully passes an SBT. SBTs are performed daily during the weaning phase, along with measurement of PiMax with airway occlusion maneuvers. Patients will be managed in a PS/CPAP mode of ventilation and PRP will be monitored continuously, adjusting PS (to a max of 20 cmH20) every 4 h to maintain PRP in the target range. PEEP may be adjusted between 5 and 10 cmH20. Weaning phase intervention continues until extubation.
- Weaning: Control: The weaning phase is defined as the time from the first SBT until the patient successfully passes an SBT. SBTs are performed daily during the weaning phase, along with measurement of PiMax with airway occlusion maneuvers. Ventilator management will be per usual care as determined by the treating clinical team until the patient is extubated.
Period: Acute Phase (0 to 28 Days)
Arm/Group | Acute: REDvent | Acute: Control | Weaning: Redvent | Weaning: Control
Started | 126 | 122 | 0 | 0
Exited Study at Acute Phase | 75 | 56 | 0 | 0
Completed | 50 | 66 | 0 | 0
Not Completed | 76 | 56 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Completed study at acute phase. | 75 | 56 | 0 | 0
Period: Weaning Phase (0 to 28 Days)
Arm/Group | Acute: REDvent | Acute: Control | Weaning: Redvent | Weaning: Control
Started (Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.) | 0 | 0 (Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.) | 58 | 58
Completed | 0 | 0 | 58 | 58
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients at baseline started in Acute: REDvent and Acute: Control arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute: REDvent | Acute: Control | Weaning: Redvent | Weaning: Control | Total
Number analyzed (Participants) | 125 | 122 | 0 | 0 | 247
Age, Categorical [Count of Participants; unit: Participants] — Population: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
  Participants
    Acute Phase Randomization: <=18 years | 120 | 117 | 0 | 0 | 237
    Acute Phase Randomization: Between 18 and 65 years | 5 | 5 | 0 | 0 | 10
    Acute Phase Randomization: >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
  years
    Acute Phase Randomization | 5.9 [1.6 to 13] | 4.9 [1.4 to 13.2] |  |  | 5.6 [1.5 to 13.1]
Age, Customized [Count of Participants; unit: Participants] — Age categories:
  infants 30 days to 365 days. Child greater than 1 year to less than 9 years Adolescents greater than or equal to 9 years Population: Measure Analysis Population Description: Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
  Participants
    Acute Phase Randomization: Infant | 20 | 21 | 0 | 0 | 41
    Acute Phase Randomization: Child | 60 | 59 | 0 | 0 | 119
    Acute Phase Randomization: Adolescents | 45 | 42 | 0 | 0 | 87
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
  Participants
    Acute Phase Randomization: Female | 54 | 61 | 0 | 0 | 115
    Acute Phase Randomization: Male | 71 | 61 | 0 | 0 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
  Participants
    Acute Phase Randomization: Hispanic or Latino | 72 | 84 | 0 | 0 | 156
    Acute Phase Randomization: Not Hispanic or Latino | 43 | 32 | 0 | 0 | 75
    Acute Phase Randomization: Unknown or Not Reported | 10 | 6 | 0 | 0 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
  Participants
    Acute Phase Randomization: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Acute Phase Randomization: Asian | 8 | 3 | 0 | 0 | 11
    Acute Phase Randomization: Native Hawaiian or Other Pacific Islander | 1 | 5 | 0 | 0 | 6
    Acute Phase Randomization: Black or African American | 11 | 8 | 0 | 0 | 19
    Acute Phase Randomization: White | 32 | 24 | 0 | 0 | 56
    Acute Phase Randomization: More than one race | 1 | 2 | 0 | 0 | 3
    Acute Phase Randomization: Unknown or Not Reported | 72 | 80 | 0 | 0 | 152
Region of Enrollment [Number; unit: participants]
  United States | 125 | 122 |  |  | 247
Number of Participants with Immunosuppression [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
  Participants | 35 | 33 | 0 | 0 | 68

OUTCOME MEASURES:

1. Primary Outcome: Median Duration of Weaning
Description: Time from first attempted SBT until SBT passage or extubation [whichever comes first]
Time Frame: First 28 days of Mechanical Ventilation
Population: Measure Analysis Population Description: All patients entered acute phase of study (n=247). Patients were eligible for the primary outcome of length of weaning if they had a spontaneous breathing trial attempted (n=215). Patients that passed first spontaneous breathing trial or were extubated successfully ended the study at the acute phase (n=131). This left 116 patients who were randomized to the weaning phase intervention.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Acute: REDvent | Acute: Control
Number analyzed (Participants) | 109 | 106
days
  Acute | 0.09 [0.08 to 2.03] | 1.04 [0.08 to 2.17]
  Weaning: number analyzed (Participants) | 56 | 58
  Weaning | 2.03 [1.09 to 3.58] | 2.10 [1.08 to 4.05]
Statistical Analysis 1: Comparison: Acute: REDvent vs Acute: Control; This analysis is comparing length of weaning between REDvent acute group and control acute group; Test type: Superiority; p = .045, Proportional Odds Logistic Regression; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.01 to 2.77]
Statistical Analysis 2: Comparison: Acute: REDvent vs Acute: Control; Weaning Phase; Test type: Superiority; Proportional odds logistic regression = 1.3, 95% CI 2-sided [0.7 to 2.6]

2. Secondary Outcome: Median Ventilator Free Days Between Acute Phase Randomization Groups
Description: Days alive and not on mechanical ventilation
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Acute: REDvent | Acute: Control
Number analyzed (Participants) | 125 | 122
days | 21.9 [14.0 to 24.5] | 21.3 [14.2 to 23.9]
Statistical Analysis 1: Comparison: Acute: REDvent vs Acute: Control; Test type: Superiority; Incident rate ratio = 1.03, 95% CI 2-sided [0.84 to 1.25] — Negative binomial model

3. Secondary Outcome: Number of Participants With Extubation Failure
Description: re-intubation
Time Frame: Within 48 hours of extubation, assessed through study completion up to maximum of 90 Days
Population: Measure Analysis Population Description: All patients entered acute phase of study (n=247). 215 patients were eligible for this outcome analysis (because they had an spontaneous breathing trial attempt.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute: REDvent | Acute: Control
Number analyzed (Participants) | 109 | 106
Participants | 8 | 8
Statistical Analysis 1: Comparison: Acute: REDvent vs Acute: Control; Test type: Superiority; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.4 to 2.7]

4. Secondary Outcome: Number of Participants With Mortality
Description: Death
Time Frame: Through study completion up to maximum of 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Acute: REDvent | Acute: Control
Number analyzed (Participants) | 125 | 122
Participants | 21 | 18
Statistical Analysis 1: Comparison: Acute: REDvent vs Acute: Control; Test type: Superiority; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.44 to 2.47]

5. Secondary Outcome: Median Maximal Inspiratory Airway Pressure During Airway Occlusion (aPiMax) at First Spontaneous Breathing Trial During Acute Phase.
Description: Measured during standardized airway occlusion maneuvers
Time Frame: Assessed on the day of first spontaneous breathing trial up to 28 days
Measure: Median (Inter-Quartile Range); unit: centimeters of water
Arm/Group | Acute: REDvent | Acute: Control
Number analyzed (Participants) | 110 | 107
centimeters of water | 51.3 [36.7 to 65] | 44.0 [34 to 60]
Statistical Analysis 1: Comparison: Acute: REDvent vs Acute: Control; Test type: Superiority; Proportional odds logistic regression = 1.60, 95% CI 2-sided [1.01 to 2.55]

6. Secondary Outcome: Median Maximal Inspiratory Esophageal Pressure During Airway Occlusion (ePiMax) During Acute Phase.
Description: Measured during standardized airway occlusion maneuvers
Time Frame: Assessed on the day of first spontaneous breathing trial up to 28 days
Measure: Median (Inter-Quartile Range); unit: centimeters of water
Arm/Group | Acute: REDvent | Acute: Control
Number analyzed (Participants) | 104 | 106
centimeters of water | 41.09 [27.5 to 52.17] | 35.5 [26.1 to 49.0]

7. Secondary Outcome: Median Percentage Change in Diaphragm Thickness on Exhalation (Dte) From Baseline During Acute Phase
Description: From daily ultrasound measurement
Time Frame: Each day from study initiation until extubation up to a maximum of 28 days
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Acute: REDvent | Acute: Control
Number analyzed (Participants) | 89 | 83
Percentage | -2 [-25 to 14] | -1 [-18 to 17]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Acute: REDvent | Acute: Control | Weaning: REDvent | Weaning: Control
All-Cause Mortality (participants affected / at risk) | 16/125 | 14/122 | 4/58 | 5/58
Serious Adverse Events (participants affected / at risk) | 19/125 | 17/122 | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 18/125 | 19/122 | 4/58 | 7/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute: REDvent (N=125) | Acute: Control (N=122) | Weaning: REDvent (N=58) | Weaning: Control (N=58)
Sustained hypoxemia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) — SpO2 less than 80% for 2 min
Air leak (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) — pneumothorax
Unplanned Extubation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial event/hemorrhage (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest/ECMO (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Progressive multi-organ failure (General disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Progression of underlying neurologic disease (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Refractory shock (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Refractory brain tumor and hypoxemia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Acute: REDvent (N=125) | Acute: Control (N=122) | Weaning: REDvent (N=58) | Weaning: Control (N=58)
Air leak (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — pneumothorax
Esphageal catheter in trachea-bronchial tree (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Failure of weaning phase (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0) — resumption of acute phase ventilation
Re-intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — within 24 hours of extubation
Sustained hypoxemia (Respiratory, thoracic and mediastinal disorders) | 12 (30) | 15 (76) | 0 (0) | 5 (6) — SpO2 less than 80% for 2 min
Unplanned Extubation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Esophageal catheter complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 1 (1) — Replacement/balloon leak/repair/agitation
Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Supra ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The structure of the trial was as described but the analytic approach was not to treat them as 4 different groups. All patients who were exposed to REDVent versus usual care during the acute phase were analyzed for outcomes attributed to the acute phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03266016/Prot_SAP_000.pdf